CLINICAL TRIAL: NCT06938880
Title: A Phase I/II Study to Evaluate the Safety, Pharmacokinetics, and Preliminary Efficacy of ZGGS18 in Combination With ZG005 in Patients With Advanced Solid Tumors, Including Cervical Cancer, Hepatocellular Carcinoma, Neuroendocrine Tumors, and Lung Cancer
Brief Title: Study of ZGGS18 in Combination With ZG005 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZGGS18-ZG005-001
Record Dates: First submitted 2025-04-07; First posted 2025-04-22 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-04

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 Dose Escalation (Experimental): ZG005 will be given 10mg/kg or 20mg/kg or other dose every three weeks and ZGGS18 will be given 10 mg/kg every three weeks
  Interventions: Biological: ZGGS18 for Injection; Biological: ZG005 for Injection
- Phase 2 Dose Expansion (Experimental): ZG005 will be given RP2D every three weeks and ZGGS18 will be given 10 mg/kg every three weeks
  Interventions: Biological: ZGGS18 for Injection; Biological: ZG005 for Injection

INTERVENTIONS:
Biological: ZGGS18 for Injection — Intravenous infusion
  Other Names: ZGGS18
Biological: ZG005 for Injection — Intravenous infusion
  Other Names: ZG005

SUMMARY:
This trial is designed to assess the tolerability, safety, pharmacokinetic profile, and preliminary efficacy of the combination of ZGGS18 and ZG005 in patients with advanced solid tumors, including advanced cervical cancer, hepatocellular carcinoma, neuroendocrine cancer, and lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand this study and voluntarily sign the ICF.
* Age 18-75 years, no gender restriction.
* Patients with advanced solid tumors who have failed standard treatment or are intolerant to standard treatment, as confirmed by histopathology or cytology.

Exclusion Criteria:

* Medical history, CT scan, or MRI indicates the presence of CNS metastases.
* Other malignancies within 5 years.
* Any other reason deeming the participant unsuitable for the study, as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Dose limited toxicity(DLT) | up to 21 days
  Incidence and severity of DLT events
Adverse Event (AE) | Up to 2 years
  Abnormal changes in clinical symptoms, vital signs, physical examination, laboratory tests, electrocardiograph and other examinations.
Maximum tolerated dose(MTD) | Up to 1 years
Recommended phase II dose(RP2D) | Up to 1 years

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  Objective Response Rate as Assessed by Investigator according to RECIST v1.1
Immunogenicity | Up to 2 years
  Incidence of antidrug antibodies (ADA)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wu, Study Chair — Suzhou Zelgen Biopharmaceuticals Co.,Ltd
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China